CLINICAL TRIAL: NCT03499886
Title: Low-Dose Intravenous Ketamine Bolus Versus Conventional Technique for Reduction of Upper and Lower Extremity Fractures in Children: A Randomized Controlled Clinical Trial
Brief Title: Low-Dose Intravenous Ketamine Bolus Versus Conventional Technique
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Principal Investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 195027
Record Dates: First submitted 2018-03-15; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Procedural Sedation
MeSH Terms: interventions — Ketamine; Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Hydrochloride 50Mg/1mL (Experimental): In the intervention group, "Ketamine Hydrochloride 50Mg/1mL" was administered rapidly at a dose of 0.5 mg / kg (within 5 seconds). Patient assessment was performed before and two minutes after ketamine injection, and then every 5 minutes after the reduction of the fracture, by an anesthetist blind to the type of intervention.
  Interventions: Drug: Ketamine Hydrochloride 50Mg/1mL Solution for Injection
- Ketamine Hydrochloride 50Mg/mL (Experimental): in the control group, ketamine 1.5 mg / kg was slowly injected for 30 to 60 seconds. Patient assessment was performed before and two minutes after ketamine injection, and then every 5 minutes after the reduction of the fracture, by an anesthetist blind to the type of intervention.
  Interventions: Drug: Ketamine Hcl 50Mg/Ml Inj

INTERVENTIONS:
Drug: Ketamine Hydrochloride 50Mg/1mL Solution for Injection — In the intervention group, ketamine 1% was administered rapidly at a dose of 0.5 mg / kg (within 5 seconds), and in the control group, ketamine 1.5 mg / kg was slowly injected for 30 to 60 seconds.
  Other Names: Ketalar
  Arms: Ketamine Hydrochloride 50Mg/1mL
Drug: Ketamine Hcl 50Mg/Ml Inj — In the intervention group, ketamine 1% was administered rapidly at a dose of 0.5 mg / kg (within 5 seconds), and in the control group, ketamine 1.5 mg / kg was slowly injected for 30 to 60 seconds.
  Arms: Ketamine Hydrochloride 50Mg/mL

SUMMARY:
Abstract Background: Ketamine has been introduced as one of the most common drugs, administered to sedate children for different painful procedures in the emergency department (ED) but administration in higher dosage causes some severe complications. Thus, the aim of this study was to evaluate the effect of low-dose intravenous ketamine bolus versus conventional injection for reduction of upper and lower extremity fractures in children.

Materials and Methods: In this randomized clinical trial, 198 participants with upper and lower extremity fractures were enrolled. The participants were divided randomly into two groups. In the intervention group, ketamine 1% was administered rapidly at a dose of 0.5 mg / kg (within 5 seconds), and in the control group, ketamine 1.5 mg / kg was slowly injected for 30 to 60 seconds. Then outcomes such as sedation depth and complications were measured for every two minutes and satisfaction of participants and physicians were recorded.

Results: Results showed that the successful sedation rate in the low dose ketamine group was significantly lower, as compared to the control group (7% vs 100%) (p<0.001). Moreover, In terms of duration of drug effect and of recovery, the low dose ketamine group were significantly lower compared with the group receiving higher dosage of ketamine (p<0.05). Furthermore, the sedation depth based on Wisconsin Sedation Scale was significantly higher, in the low dose ketamine group compared to the other group. By evaluating different complications, we found that the rate of neurological (20.4 % vs 5%) and physiological (10.2% vs 2%) complications in the control group was significantly higher compared to the group receiving low-dose ketamine (p<0.05).

DETAILED DESCRIPTION:
This prospective double-blind clinical trial was conducted in the ED of Isfahan Al-Zahra Hospital, from May 2016 to June 2017. The sedation levels and different outcomes of patients receiving low-dose intravenous ketamine bolus (intervention group) were compared to patients receiving higher doses of intravenous ketamine (control group), for reduction of upper and lower extremity fractures. Inclusion criteria consisted of parents' desire and consent to participate in the study, body mass index (BMI) within the normal range, having age of 6 months to 17 years, requiring a reduction of upper and lower limb fractures, not receiving benzodiazepines and other sedative drugs before intervention.

Exclusion criteria consisted of patients' age <3 months with the body temperature of > 38 ̊C, due to upper respiratory tract infection. Patients having any other complications such as cardiovascular, gastrointestinal, psychological and neurological were excluded from the study. We also excluded the patients who have withdrawn from the study.

Participants and Intervention The study flowchart is shown in figure 1. Two hundreds ten patients with a diagnosis of upper and lower extremity fractures, diagnosed by Emergency Medicine Specialist, were enrolled based on clinical and para-clinical images and inclusion criteria.

The participants were randomly allocated into two groups, using a block randomization procedure with matching subjects in each block based on sex and age. One hundred ninety eight patients completed the study; including one hundred from the intervention group and 98 from the control group. The study received ethics approval from the Ethics Committee of Isfahan University of Medical Sciences (--------------), and all participants and their parents signed the informed consent form.

After obtaining informed consent, eligible patients were enrolled. All patients were monitored by direct observation and continuous cardiovascular monitoring, in order to check the vital signs and also by pulse Oximeters to examine the blood oxygen saturation level.

ELIGIBILITY:
Inclusion Criteria:

* Parents' desire and consent to participate in the study
* Body mass index (BMI) within the normal range
* Having age of 6 months to 17 years
* Requiring a reduction of upper and lower limb fractures.
* Subjects who did not complete study endpoints, however, were included as part on an intention to treat analysis.

Exclusion Criteria:

* Age <6 months
* Body temperature of > 38 ̊C, due to upper respiratory tract infection.
* Participants having any other complications such as cardiovascular, gastrointestinal, psychological and neurological .
* Patients who have withdrawn from the study, or those receiving benzodiazepines and other sedative drugs within 6 hours prior to enrollment.
* Subjects who refused to give consent or those who were judged by investigator as non eligible were excluded as well.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 198 (Estimated)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-04-28 (Estimated); Study Completion 2018-05-14 (Estimated)

PRIMARY OUTCOMES:
Sedation depth | 30 minutes
  By Ramsey sedation scale. With score 1 for restlessness to score 6 for unresponsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Nasr Isfahani, M.D., Principal Investigator — Isfahan University of Medical Sciences
Locations (2):
- Iran (2):
  - Al-Zahra University Hospital, Isfahan
  - Mehdi Nasr Isfahani, Isfahan

IPD SHARING:
Plan to Share IPD: Undecided